CLINICAL TRIAL: NCT02460289
Title: Multicenter, Open Label Clinical Trial to Evaluate the Effect and Tolerability of Minoxidil 5% Foam and Botanical Hair Solution Regimen in Men With Thinning Hair and Male Pattern of Hair Loss/Androgenic Alopecia (Norwood III & IV)
Brief Title: Minoxidil 5% / Botanical Hair Regimen in Men With Thinning Hair and Male Pattern Hair Loss/Androgenic Alopecia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.SPR.US 10329
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Male Pattern of Hair Loss, Androgenic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Menogaril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Treatment: Minoxidil 5% / Botanical Hair Solution for Men

INTERVENTIONS:
Drug: Treatment: Minoxidil 5% / Botanical Hair Solution for Men

SUMMARY:
The purpose of this study is to characterize the effect of Minoxidil 5% Foam and Botanical Hair Solution Regimen in men with thinning hair and male pattern hair loss/androgenic alopecia (Norwood III & IV).

ELIGIBILITY:
Key Inclusion Criteria:

1. Male patients age 18 to 60 years at the time of enrollment.
2. Men who have self-perceived thinning hair.
3. Men who have presentation of male pattern hair loss/androgenic alopecia (Norwood III & IV).

Key Exclusion Criteria:

1. History of allergic reactions or severe intolerance to minoxidil and Botanical Hair Solution product ingredients.
2. Plan to use any other concomitant therapy to treat hair loss, regrowth or volume during the study.

3 Subjects taking or planning to take topical or systemic prescription or OTC medications for treating hair loss and/or hair volume.

4. Any significant history of concurrent medical disease, which in the judgment of the Investigator, would make the subject inappropriate for entry to this study including history of skin disease that may confound study results.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2015-05-19 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren Winkelman, MD, PhD, MBA, Study Director — Galderma R&D
Locations (1):
- Stephens & Associates, Richardson, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in the United States from 19 May 2015 to 19 September 2015.
Groups:
- Minoxidil 5% Foam and Botanical Hair Solution for Men: Participant were applied with minoxidil 5% foam on the scalp in the hair loss and botanical hair solution (5-10 sprays) for men on entire scalp (wet or dry) twice per day for 12 weeks.
Period: Overall Study
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution for Men
Started | 63
Intent to Treat (ITT) Population | 56
Safety Population (SP) | 61
Completed | 53
Not Completed | 10
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: SP included all participants who were enrolled and received at least one dose of study product.
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution for Men
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 4
  Black or African American | 6
  Hispanic or Latino | 11
  White | 37
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick skin type is a numerical classification scale for the color of skin from Type 1 to Type VI. I - Always bums; never tans II - Bums easily; tans minimally III - Burns moderately; tans gradually to light brown IV - Burns minimally; tans well to moderate brown V - Rarely burns; tans profusely to dark brown VI - Never bums; tans profusely to black.
  Participants
    II | 6
    III | 32
    IV | 18
    V | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Investigator's Rating of Standardized Global Photographs at Week 12
Description: The Investigator or a trained grader rated each participant's standardized global photographs for improvement from baseline for parameters like hair thinning, hair growth, impression of scalp hair coverage and overall perception of treatment benefit using a 1-to-7-point Likert scale. Investigator global photograph rating were assessed using 7-point Likert scale. Each score on the individual scale ranged from 1 (minimum) to 7 (maximum), that is, (1) Entirely Disagree; (2) Mostly Disagree; (3) Somewhat Disagree; (4) Neither Agree nor Disagree; (5) Somewhat Agree; (6) Mostly Agree; (7) Entirely Agree.
Time Frame: At Week 12
Population: ITT population included all participants who were randomized and have at least one post-treatment administration evaluation.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution for Men
Number analyzed (Participants) | 56
Score on a scale
  Hair Thinning | 5.0 (0.9)
  Hair Growth | 5.1 (0.9)
  Impression of scalp hair coverage | 5.1 (0.9)
  Overall perception of treatment benefit | 5.1 (0.9)

2. Primary Outcome: Change From Baseline in Participant Rating at Week 12
Description: Participants rated the parameters like appearance of hair, growth of hair, satisfaction with hairline at the front of the head, satisfaction with hair on the top of the head and satisfaction with hair overall as an overall improvement from the baseline by conducting their own assessments by looking in a mirror and evaluating improvement from baseline using a 1 to 7-point Likert scale. Each score on the individual scale ranged from 1 (minimum) to 7 (maximum), that is, (1) Entirely Disagree; (2) Mostly Disagree; (3) Somewhat Disagree; (4) Neither Agree nor Disagree; (5) Somewhat Agree; (6) Mostly Agree; (7) Entirely Agree.
Time Frame: At Week 12
Population: lIT population included all participants who were randomized and had at least one post-treatment administration evaluation.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution for Men
Number analyzed (Participants) | 56
Score on a scale
  Appearance of hair | 5.4 (1.2)
  Growth of hair | 5.3 (1.3)
  Satisfaction with hairline at the front of the head | 4.9 (1.4)
  Satisfaction with hair on the top of the head | 5.0 (1.5)
  Satisfaction with hair overall as an overall improvement | 5.2 (1.4)

3. Secondary Outcome: Mean Change From Baseline in Shed Hair Count
Description: Participants collected their hair full day, including after combing and hair-washing. Participants turned in these hair collections at each visit. The results were averaged weekly. Mean change from baseline in hair wash/shed hair count was reported at Week 12.
Time Frame: At Week 12
Population: lTT population included all participants who were randomized and had at least one post-treatment administration evaluation.
Measure: Mean (Standard Deviation); unit: Shed Hair Count
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution for Men
Number analyzed (Participants) | 56
Shed Hair Count | 14.1 (21.6)

4. Secondary Outcome: Number of Participant in Each Response Category Based on Subject Satisfaction Questionnaire
Description: Participant's satisfaction questionnaire was used to specifically collect the participants' feedback on the treatment regimen, the level of satisfaction and future usage. Participants were asked to complete a cosmetic acceptability questionnaire. This 10 item questionnaire had a 5-point Likert Response Scale (1=Strongly Agree; 5=Strongly Disagree).
Time Frame: At Week 4,6 and 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution for Men
Number analyzed (Participants) | 56
Participants
  Satisfaction with appearance of hair (At Week 4): Agree | 27
  Satisfaction with appearance of hair (At Week 4): Disagree | 8
  Satisfaction with appearance of hair (At Week 4): Neutral | 21
  Satisfaction with appearance of hair (At Week 6): Agree | 42
  Satisfaction with appearance of hair (At Week 6): Disagree | 4
  Satisfaction with appearance of hair (At Week 6): Neutral | 10
  Satisfaction with appearance of hair (At Week 12): Agree | 44
  Satisfaction with appearance of hair (At Week 12): Disagree | 4
  Satisfaction with appearance of hair (At Week 12): Neutral | 8
  Satisfaction with growth of hair (At Week 4): Agree | 26
  Satisfaction with growth of hair (At Week 4): Disagree | 12
  Satisfaction with growth of hair (At Week 4): Neutral | 18
  Satisfaction with growth of hair (At Week 6): Agree | 40
  Satisfaction with growth of hair (At Week 6): Disagree | 5
  Satisfaction with growth of hair (At Week 6): Neutral | 11
  Satisfaction with growth of hair (At Week 12): Agree | 44
  Satisfaction with growth of hair (At Week 12): Disagree | 7
  Satisfaction with growth of hair (At Week 12): Neutral | 5
  Satisfaction with hairline at the front of the head (At Week 4): Agree | 21
  Satisfaction with hairline at the front of the head (At Week 4): Disagree | 16
  Satisfaction with hairline at the front of the head (At Week 4): Neutral | 19
  Satisfaction with hairline at the front of the head (At Week 6): Agree | 26
  Satisfaction with hairline at the front of the head (At Week 6): Disagree | 10
  Satisfaction with hairline at the front of the head (At Week 6): Neutral | 20
  Satisfaction with hairline at the front of the head (At Week 12): Agree | 34
  Satisfaction with hairline at the front of the head (At Week 12): Disagree | 8
  Satisfaction with hairline at the front of the head (At Week 12): Neutral | 14
  Satisfaction with hair on the top of the head (At Week 4): Agree | 21
  Satisfaction with hair on the top of the head (At Week 4): Disagree | 16
  Satisfaction with hair on the top of the head (At Week 4): Neutral | 19
  Satisfaction with hair on the top of the head (At Week 6): Agree | 36
  Satisfaction with hair on the top of the head (At Week 6): Disagree | 7
  Satisfaction with hair on the top of the head (At Week 6): Neutral | 13
  Satisfaction with hair on the top of the head (At Week 12): Agree | 37
  Satisfaction with hair on the top of the head (At Week 12): Disagree | 7
  Satisfaction with hair on the top of the head (At Week 12): Neutral | 12
  Satisfaction with hair overall as an overall improvement from the baseline (At Week 4): Agree | 21
  Satisfaction with hair overall as an overall improvement from the baseline (At Week 4): Disagree | 13
  Satisfaction with hair overall as an overall improvement from the baseline (At Week 4): Neutral | 22
  Satisfaction with hair overall as an overall improvement from the baseline (At Week 6): Agree | 34
  Satisfaction with hair overall as an overall improvement from the baseline (At Week 6): Disagree | 5
  Satisfaction with hair overall as an overall improvement from the baseline (At Week 6): Neutral | 17
  Satisfaction with hair overall as an overall improvement from the baseline (At Week 12): Agree | 39
  Satisfaction with hair overall as an overall improvement from the baseline (At Week 12): Disagree | 6
  Satisfaction with hair overall as an overall improvement from the baseline (At Week 12): Neutral | 11

5. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs)
Description: AEs were defined as any untoward medical occurrence associated with the use of a study product in humans, whether or not considered study product related. An AE could be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study product and would not imply any judgment about causality. An AE could arise with any use of the study product and with any route of administration, formulation, or dose, including an overdose. Thus, any new sign, symptom or disease, or clinically significant increase in the intensity of an existing sign, or symptom would be considered as an AE. Any new clinically relevant sign or symptom suffered by the participant, which appeared after the study procedures was reported as an AE. Any worsening in scalp dryness or itch score from baseline was also reported as an AE. The Investigator or designee had the final authorization to determine if a reaction was considered an AE.
Time Frame: From start of study up to Week 12
Population: SP included all participants who were enrolled and received at least one dose of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution for Men
Number analyzed (Participants) | 61
Participants | 4

ADVERSE EVENTS:
Time Frame: From Start of Study up to Week 12
Description: The safety population was defined as all participants who were enrolled and received at least one dose of study product.
Arm/Group | Minoxidil 5% Foam and Botanical Hair Solution for Men
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 4/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Minoxidil 5% Foam and Botanical Hair Solution for Men (N=61)
Pain (crown of head) (General disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Joint Injury (Musculoskeletal and connective tissue disorders) | 1
Middle ear effusion (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes